CLINICAL TRIAL: NCT04534569
Title: Expert Panel Statement for the Respiratory Management of COVID-19 Related Acute Respiratory Failure (C-ARF) Using Modified Delphi Methodology
Brief Title: Expert Panel Statement for the Respiratory Management of COVID-19 Related Acute Respiratory Failure (C-ARF)
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Responsible Party: Principal Investigator, Prashant Nasa, Head Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: C19ARFstudy
Record Dates: First submitted 2020-08-30; First posted 2020-09-01 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Acute Respiratory Failure; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Experts consensus — Consensus opinion using Delphi Methodology

SUMMARY:
The investigators aim to achieve experts consensus on respiratory interventions in management of COVID-19 related acute respiratory failure (C-ARF).

DETAILED DESCRIPTION:
The investigators aim to achieve experts consensus on respiratory interventions in management of COVID-19 related acute respiratory failure (C-ARF). The pandemic of COVID-19 is unique in terms of a multitude of patients suffering from ARF and requiring invasive mechanical ventilation with single underlying inciting etiology.The experts have given divergent opinions on respiratory support of C-ARF which may have confused physicians globally.

The investigators are going to use a modified Delphi based methodology involving global participating experts. The objective is to achieve consensus statement on the management of C-ARF using "collective intelligence".

The whole process of this study will be done in the form of two-three rounds of Google Forms-based Delphi surveys. In this survey questionnaire, the investigators have prepared statements on the concern areas in the respiratory support of C-ARF. The survey has been divided into five sections related to C-ARF management. The majority of these statements are to be rated on Likert scale and others have multiple choices. There is an option for collecting participating experts comments in provided open space in round one which will be considered during round two questionnaire.

ELIGIBILITY:
Inclusion Criteria: (All the three criteria should be there) H index more than 10; one or more publication on respiratory failure in indexed journal; actively involved in management of COVID-19 related acute respiratory failure.

Exclusion Criteria:

Not meeting inclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Global Experts in Respiratory or Critical Care Medicine
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Consensus using participating experts opinions. | 20 days
  Survey Questionnaire containing seven point Likert scale and multiple choice questions.

CONTACTS AND LOCATIONS:
Locations (1):
- NMC Specialty Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narendra DK, Hess DR, Sessler CN, Belete HM, Guntupalli KK, Khusid F, Carpati CM, Astiz ME, Raoof S. Update in Management of Severe Hypoxemic Respiratory Failure. Chest. 2017 Oct;152(4):867-879. doi: 10.1016/j.chest.2017.06.039. Epub 2017 Jul 14. PMID 28716645
- [Background] Tang S, Mao Y, Jones RM, Tan Q, Ji JS, Li N, Shen J, Lv Y, Pan L, Ding P, Wang X, Wang Y, MacIntyre CR, Shi X. Aerosol transmission of SARS-CoV-2? Evidence, prevention and control. Environ Int. 2020 Nov;144:106039. doi: 10.1016/j.envint.2020.106039. Epub 2020 Aug 7. PMID 32822927
- [Derived] Nasa P, Azoulay E, Khanna AK, Jain R, Gupta S, Javeri Y, Juneja D, Rangappa P, Sundararajan K, Alhazzani W, Antonelli M, Arabi YM, Bakker J, Brochard LJ, Deane AM, Du B, Einav S, Esteban A, Gajic O, Galvagno SM Jr, Guerin C, Jaber S, Khilnani GC, Koh Y, Lascarrou JB, Machado FR, Malbrain MLNG, Mancebo J, McCurdy MT, McGrath BA, Mehta S, Mekontso-Dessap A, Mer M, Nurok M, Park PK, Pelosi P, Peter JV, Phua J, Pilcher DV, Piquilloud L, Schellongowski P, Schultz MJ, Shankar-Hari M, Singh S, Sorbello M, Tiruvoipati R, Udy AA, Welte T, Myatra SN. Expert consensus statements for the management of COVID-19-related acute respiratory failure using a Delphi method. Crit Care. 2021 Mar 16;25(1):106. doi: 10.1186/s13054-021-03491-y. PMID 33726819